CLINICAL TRIAL: NCT07225530
Title: Implementation of Screen, Treat, and Triage for Women Living With HIV in La Romana (iSTAR)
Acronym: (iSTAR)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Clínica de Familia La Romana, Dominican Republic (Unknown)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AAAV3441; U01CA275110 (NIH)
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections; HPV Infection; Cervical Cancer
Keywords: People living with HIV (PLWH); Cervical cancer screening; Spanish speakers; HPV Infection
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Mass Screening; Triage; Coal Tar

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of two trial arms through REDCap using randomly permuted block design where the block size itself is randomly selected, treatment assignment is pre-determined before the trial begins, and assignments remain static throughout the course of the trial to reduce opportunities for selection bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants randomized to the standard of care group will receive standard examinations and management of screen positives (ablative therapy or colposcopy referral at a follow-up visit).
- Screen, Triage, and Treat (Experimental): Participants randomized to the screen, triage, and treat group will be examined using the screen and treat approach (same day results and ablative therapy or colposcopy referral, if applicable).
  Interventions: Other: Screen, Triage, and Treat

INTERVENTIONS:
Other: Screen, Triage, and Treat — A screening test is used to determine who is eligible for treatment, eliminating steps related to histological confirmation. Those who meet the HPV criteria will be immediately evaluated for suitability for on-site ablative treatment on the same day. Women not suitable for treatment will be referred for colposcopy and further management at the appropriate facility.
  Arms: Screen, Triage, and Treat

SUMMARY:
This study aims to conduct a randomized controlled trial to evaluate the effectiveness of same-day HPV-based screen and treat among women living with HIV (WLH) in La Romana, Dominican Republic. With cervical cancer being a leading cause of cancer-related deaths in women living with HIV, and cervical cancer deaths being preventable through screening and early detection, this project seeks to identify factors associated with the successful implementation of the Screen, Triage, and Treat approach to inform future implementation and scale-up.

DETAILED DESCRIPTION:
The Dominican Republic (DR) has experienced a high burden of human immunodeficiency virus (HIV) over the last two decades. Unlike the United States, women are represented in almost equal numbers to men in the population living with HIV. Cervical cancer is the most common cancer among Women Living with HIV (WLH) and WLH are more likely to be infected with HPV and have persistent human papillomavirus (HPV) infection leading to precancer. Additionally, Latin America and the Caribbean are second only to sub-Saharan Africa in their cervical cancer burden. The DR has both a higher incidence of cervical cancer and a higher mortality rate from cervical cancer than the rest of the Caribbean. In fact, cervical cancer is the leading cause of cancer death for women 15-44 years of age in the DR. Cervical cancer persists in the DR largely because of the failure of routine screening. Coverage for cervical cancer screening is less than 50%, and fewer than 25% of the screen-positives complete the full round of follow-up care. Screening programs are critical so that every woman with precursor lesions is treated, and avoidable deaths are prevented. For a cervical cancer prevention and control program to have impact, retention in a full cycle of screening and treatment is fundamental.

The purpose of this randomized clinical trial (RCT) is to evaluate, through use of a clinical decision support system (CDSS), the effectiveness of primary screening for HPV using either the iSTAR approach with same day results return and same-day treatment for those eligible compared to standard of care (SOC). The iSTAR approach circumvents the multistep screening process by conducting the screening test (HPV), the triage step (HPV VL), and if suitable for ablative therapy, the treatment procedure (thermocoagulation) in a single visit. Those who are HPV positive and meet the HPV VL triage criteria but are not suitable for ablative therapy (large lesions, upper limit not seen, etc.) are referred to colposcopy services. This study will allow us to evaluate potential strategies for ensuring widespread implementation of Screen, Triage, and Treat in future work.

ELIGIBILITY:
Inclusion Criteria:

* 25 years of age;
* female sex assigned at birth (any gender identity);
* HIV-positive;
* women who have had cervical cancer precursor lesions which were removed more than 6 months ago; and
* understand Spanish

Exclusion Criteria:

* ages outside of the specified inclusion criteria;
* women who are pregnant, less than 6 weeks postpartum, or in whom pregnancy cannot be excluded;
* history of a Loop Electrosurgical Excision Procedure (LEEP) procedure in the last 6 months;
* history of a hysterectomy;
* previous diagnosis of gynecological cancer;
* history of cancer of the anogenital tract; or
* unable or unwilling to provide informed consent

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Screen-positives Completing Full Screening Cascade | 2 Months
  The investigators will calculate the percent of screen-positives who complete all follow-up steps in the screening cascade. For the iSTAR approach, this will include the percentage among those suitable for ablative therapy who undergo ablative therapy within 1 week of screening combined with the percentage of those not suitable for ablative therapy who complete all colposcopy referral steps which lead either to a treatment procedure or to a negative confirmatory diagnosis within 2 months. In the standard of care arm, this will include the percentage of all screen-positives who complete the colposcopy steps within 2 months.
Percentage of Women in the HPV+VL Triage Negative Group | Day 1
  The investigators will calculate the percentage of women with HPV+ by HPV VL triage negative who have abnormal pap results. Given the high specificity of cytology, this will quantify the extent of missed disease with the HPV VL triage approach.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, Principal Investigator — Columbia University
Locations (1):
- Clínica de Familia La Romana, La Romana, Dominican Republic

IPD SHARING:
Plan to Share IPD: No